CLINICAL TRIAL: NCT02040259
Title: Stryker Neurovascular Trevo® Retriever Registry
Brief Title: Trevo® Retriever Registry Post Market Surveillance
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: T4025
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; mechanical thrombectomy device; Retriever
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical thrombectomy, Trevo Retriever: Mechanical thrombectomy, Trevo Retriever

SUMMARY:
The purpose of the Trevo® Retriever Registry is to collect real world performance data of the Trevo Retriever which is intended to restore blood flow in the neurovasculature by removing thrombus in patients experiencing ischemic stroke.

DETAILED DESCRIPTION:
Trevo Retriever Registry is a prospective, open-label, consecutive enrollment, multi-center, international registry that may enroll a maximum of 2000 patients at up to 100 sites worldwide. Revascularization status will be assessed at the end of the procedure using the modified TICI (Thrombolysis in Cerebral Infarction)score. Additional data collection will include:

1. Day 90 mRS assessment
2. Day 90 all cause mortality
3. Neurological deterioration at 24 hours post procedure, defined as a four or more point increase in the NIHSS score from the baseline score
4. Rates of device and procedure related serious adverse events (AEs)

ELIGIBILITY:
Inclusion Criteria:

* Subjects experiencing acute ischemic stroke who are eligible for restoration of blood flow using any approved Trevo Retriever in the neurovasculature to remove thrombus
* Trevo Retriever is the initial mechanical neuro-thrombectomy device used to remove the thrombus
* Signed Informed Consent obtained
* Subject willing to comply with the protocol follow-up requirements
* Anticipated life expectancy of at least 3 months

Exclusion Criteria:

* The subject is participating in another mechanical neuro-thrombectomy device trial or any other clinical trial where the study procedure or treatment might confound the study end point.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute ischemic stroke patients who may be referred for mechanical thrombectomy is used to removed thrombus in the neurovasculature
Sampling Method: Probability Sample
Enrollment: 2008 (Actual)
Dates: Start 2013-11-25; Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Veznedaroglu, MD, Principal Investigator — Drexel Neurosciences Institute,Philadelphia; Ronald Budzik, MD, Principal Investigator — Riverside Methodist Hospital/ Ohio Health Research Institute, Columbus, OH
Locations (80):
- United States (47):
  - Banner Desert Medical Center, Mesa, Arizona
  - St. Joseph's Hospital and Medical Center - Dignity Health (BNI Phoenix), Phoenix, Arizona
  - Eden Medical Center, Castro Valley, California
  - St. Jude Medical Center, Fullerton, California
  - Scripps Memorial Hospital, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - UCI Medical Center, Orange, California
  - California Pacific Medical Center (CPMC), San Francisco, California
  - Good Samaritan Hospital Regional Medical Center, San Jose, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Yale University / Yale-New Haven Hospital, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist Medical Center - Jacksonville, Jacksonville, Florida
  - University of Miami (Jackson Memorial), Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Center for Advanced Research Excellence (St. Mary's Medical Center), West Palm Beach, Florida
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Advocate Christ Lutheran Hospital, Park Ridge, Illinois
  - Peoria Radiology Research & Education Foundation, Peoria, Illinois
  - University of Iowa, Iowa City, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - UMass Memorial, Worcester, Massachusetts
  - McLaren Flint Regional Medical Center, Flint, Michigan
  - St. Joseph Mercy, Pontiac, Michigan
  - Capital Health System, Trenton, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - Mount Sinai Health System, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Mission Hospital, Asheville, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital/ Ohio Health Research Institute, Columbus, Ohio
  - Oregon Stroke Center, Oregon Health & Science University (OHSU), Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Erlanger Hospital, Chattanooga, Tennessee
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - Methodist Healthcare - Memphis Hospitals, Memphis, Tennessee
  - Valley Baptist Harlingen, Harlingen, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
- Toronto Western Hospital, Toronto, Canada
- University Hospital Hradec Králové, Hradec Králové, Czechia
- France (9):
  - CHU Bordeaux, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - GRENOBLE, Grenoble
  - CHU Lille, Lille
  - Hopital Dupuytren, Limoges
  - CHU Nancy, Nancy
  - La Pitié Salpêtrière, Paris
  - La Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - CHU de Tours, Tours
- Germany (9):
  - Klinikum Augsburg, Augsburg
  - Vivantes Klinikum Neukölln, Berlin
  - Klinikum Dortmund, Dortmund
  - Uniklinik Erlangen, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Uniklinik Heidelberg, Heidelberg
  - Uniklinik Homburg, Homburg/ Saar
  - UKSH; Lübeck, Lübeck
  - Uniklinik Mainz- Mainz, Mainz-GE
- National Institute of Clinical Neurosciences, Budapest, Hungary
- Italy (2):
  - Spedali Civili di Brescia, Brescia
  - Ospedale San Martino, Genova
- National Neuroscience Institute,, Singapore, Singapore
- South Korea (2):
  - Kyungpook National University Hospital, Jungni I Gu
  - Seoul National University Bundang Hospital, Seongnam-si
- Spain (5):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
  - Son Espases de Mallorca, Palma de Mallorca
- Kantonsspital Aarau, Aarau, Switzerland
- Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Bartolini B, Krajina A, Budzik R, Gupta R, Nogueira RG, Malek A, Sarraj A, English J, Narata AP, Taqi M, Miller T, Grobelny T, Baxter B, Jenkins P, Liebeskind DS, Veznedaroglu E; Trevo Registry Investigators. Outcomes of Mechanical Thrombectomy of Acute Basilar Artery Occlusion Due to Underlying Intracranial Atherosclerotic Disease. Stroke Vasc Interv Neurol. 2022 Nov 18;3(2):e000429. doi: 10.1161/SVIN.122.000429. eCollection 2023 Mar. PMID 41585922
- [Derived] Nogueira RG, Haussen DC, Liebeskind D, Jovin TG, Gupta R, Jadhav A, Budzik RF, Baxter B, Krajina A, Bonafe A, Malek A, Narata AP, Shields R, Zhang Y, Morgan P, Bartolini B, English J, Frankel MR, Veznedaroglu E; Trevo Registry and DAWN Trial Investigators. Stroke Imaging Selection Modality and Endovascular Therapy Outcomes in the Early and Extended Time Windows. Stroke. 2021 Jan;52(2):491-497. doi: 10.1161/STROKEAHA.120.031685. Epub 2021 Jan 12. PMID 33430634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Trevo Retriever Registry was a prospective, open-label, consecutive enrollment, multi-center international registry designed to enroll up to 2,000 subjects at up to 100 clinical sites worldwide.
Groups:
- Mechanical Thrombectomy, Trevo Retriever: The Trevo Retriever registry was a prospective, open-label, consecutive enrollment, multi-center global registry to assess real world performance of the Trevo Retriever which is intended to restore blood flow in the neurovasculature be removing thrombus in subjects experiencing ischemic stroke
Period: Overall Study
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
Started | 2008
Completed | 1645
Not Completed | 363
Not completed — Death | 280
Not completed — Lost to Follow-up | 76
Not completed — Assessment not completed | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Trevo Retriever: Mechanical thrombectomy, Trevo Retriever
Arm/Group | Trevo Retriever
Number analyzed (Participants) | 2008
Age, Categorical [Count of Participants; unit: Participants] — Baseline demographics included in the intent to treat population.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 735
    >=65 years | 1273
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1041
  Male | 967
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 8
  South Korea | 27
  Singapore | 8
  Hungary | 28
  United States | 1365
  Czechia | 131
  Italy | 12
  France | 183
  Thailand | 20
  Switzerland | 9
  Germany | 83
  Spain | 134

OUTCOME MEASURES:

1. Primary Outcome: Revascularization Status Assessment at the End of the Trevo Retriever Procedure Using the Modified TICI Score
Description: The primary end point is revascularization based on modified Thrombolysis in Cerebral Infarction score (mTICI). Per protocol, successful revascularization is defined as having a modified TICI score ≥2b at the end of the procedure.
  Modified TICI Scale (mTICI Scale) Grade 0 - No Perfusion Grade 1 - Penetration with Minimal Perfusion Grade 2 - Partial Perfusion Grade 2a - Only partial filling (< 50%) of the entire vascular territory is visualized.
  Grade 2b - Filling of > 50% all of the expected vascular territory is visualized, but the filling is slower than normal.
  Grade 3 - Complete Perfusion
Time Frame: Post Procedure
Population: Intention to Treat (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- Mechanical Thrombectomy, Trevo Retriever: Study participants undergoing mechanical thrombectomy, with the Trevo Retriever
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
Number analyzed (Participants) | 2008
Participants | 1863

2. Secondary Outcome: Modified Rankin Scale (mRS) Assessment at 90 Days
Description: The Modified Rankin Scale mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  A good clinical outcome = mRS scale 0-2. 0 - No symptoms at all.
  1. - No significant disability despite symptoms; able to carry out all usual duties and activities.
  2. - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance.
  3. - Moderate disability; requiring some help, but able to walk without assistance.
  4. - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance.
  5. - Severe disability; bedridden, incontinent and requiring constant nursing care and attention.
  6. - Dead.
Time Frame: 90 days
Population: Per Protocol. This endpoint includes patient with a baseline and 90 day assessment. 1997 participants that underwent mechanical thrombectomy with the Trevo retriever completed both assessments.
Measure: Count of Participants; unit: Participants
Groups:
- Mechanical Thrombectomy, Trevo Retriever: Study participants that have undergone mechanical thrombectomy with Trevo retriever with a completed modified Rankin Scale assessment at baseline and 90 days.
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
Number analyzed (Participants) | 1997
Participants | 1104

3. Secondary Outcome: All Cause Mortality
Description: Overall mortality rate
Time Frame: 90 days
Population: Intention to Treat (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- Mechanical Thrombectomy, Trevo Retriever: Study participants that have undergone mechanical thrombectomy with Trevo retriever.
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
Number analyzed (Participants) | 2008
Participants | 280

4. Secondary Outcome: Device and Procedure Related Serious Adverse Events (SAEs)
Description: Rate of Device and Procedure related serious adverse events (SAE)
Time Frame: 90 days
Population: Intention to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
Number analyzed (Participants) | 2008
Participants | 49

5. Secondary Outcome: Neurological Deterioration at 24 Hours
Description: Neurological Deterioration at 24 hours post procedure, defined as a 4 point or more increase in the NIHSS score over the baseline score.
Time Frame: 24 hours
Population: Intention to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
Number analyzed (Participants) | 2008
Participants | 97

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Mechanical Thrombectomy, Trevo Retriever
All-Cause Mortality (participants affected / at risk) | 280/2008
Serious Adverse Events (participants affected / at risk) | 427/2008
Other Adverse Events (participants affected / at risk) | 174/2008
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mechanical Thrombectomy, Trevo Retriever (N=2008)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial septal defect (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 20
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 8
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 7
Cardiac valve disease (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Cardio respiratory arrest (Cardiac disorders) | 6
Cardiopulmonary failure (Cardiac disorders) | 3
Intracardiac thrombus (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 2
Mitral valve stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 4
Sick sinus syndrome (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Intestinal ichaemia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Perirectal abscess (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Autonomic nervous system imbalance (General disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 11
Delirium tremens (General disorders) | 1
General physical health deterioration (General disorders) | 1
Multi-organ failure (General disorders) | 1
Organ failure (General disorders) | 1
Liver abscess (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Cholecystitis infective (Infections and infestations) | 1
Cholstridium difficule infection (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 17
Pseudomonal bacteraemia (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 14
Septic shock (Infections and infestations) | 7
Staphylococcal infections (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1
Complications of transplanted heart (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Traumatic intracranial hemmorrhage (Injury, poisoning and procedural complications) | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 7
Vascular pseudoneurysm (Injury, poisoning and procedural complications) | 1
Vessel perforation (Injury, poisoning and procedural complications) | 8
Haemoglobin decreased (Investigations) | 1
International normalised ratio abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gliblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mestastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basilar artery occlusion (Nervous system disorders) | 1
Brain death (Nervous system disorders) | 1
Brain herniation (Nervous system disorders) | 2
Brain oedema (Nervous system disorders) | 18
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral artery embolism (Nervous system disorders) | 3
Cerebral artery occlusion (Nervous system disorders) | 1
Cerebral artery thrombosis (Nervous system disorders) | 2
Cerebral haematoma (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral hyperperfusion syndrome (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 10
Coma (Nervous system disorders) | 1
Complex partial seizures (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 4
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Gasping syndrome (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 51
Haemorrhagic stroke (Nervous system disorders) | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 5
Neurological decompensation (Nervous system disorders) | 96
Partial seizures (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Stroke in evolution (Nervous system disorders) | 5
Transient Ischaemic attach (Nervous system disorders) | 2
Vasogenic cerebral oedema (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 11
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 27
Homicide (Social circumstances) | 1
Mitral valve replacement (Surgical and medical procedures) | 1
Artery dissection (Vascular disorders) | 3
Cardiogenic shock (Vascular disorders) | 2
Cerebral artery embolism (Vascular disorders) | 1
Cerebral artery thrombosis (Vascular disorders) | 1
Cerebral haematoma (Vascular disorders) | 1
Cerebral infarction (Vascular disorders) | 1
Coeliac artery stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Extravasation blood (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Peripheral ischaemia (Vascular disorders) | 1
Shock (Vascular disorders) | 4
Subarachnoid haemorrhage (Vascular disorders) | 2
Syncope (Vascular disorders) | 1
Vascular dissection (Vascular disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mechanical Thrombectomy, Trevo Retriever (N=2008)
Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Normachromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Atrioventricular block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pulmonary oedema (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Eye inflammation (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Extravasation (General disorders) | 1
Tobacco withdrawal symptoms (General disorders) | 1
Vessel puncture site haematoma (General disorders) | 1
Drug hypersenitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Hypersensitivity (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia pseudomonal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 14
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Vessel perforation (Injury, poisoning and procedural complications) | 5
Blood pressure increased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Magnesium metabolism disorder (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Intracranial germ cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal ganglia infarction (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebral artery embolism (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral vasoconstriction (Nervous system disorders) | 10
Cerebrovascular accident (Nervous system disorders) | 2
Confusional state (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 13
Headache (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 54
Subarachnoid haemorrhage (Nervous system disorders) | 2
Anuria (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Artery dissection (Vascular disorders) | 2
Cerebral artery embolism (Vascular disorders) | 2
Cerebral artery thrombosis (Vascular disorders) | 1
Cerebral haemorrhage (Vascular disorders) | 2
Haemorrhage intracranial (Vascular disorders) | 13
Haemorrhagic transformation stroke (Vascular disorders) | 3
Mouth haemorrhages (Vascular disorders) | 1
Subarachnoid haemorrhage (Vascular disorders) | 5
Uterine haemorrhage (Vascular disorders) | 1
Vascular dissection (Vascular disorders) | 3
Pyrexia (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician shall not make any publication without providing Sponsor 60 days notice. If Sponsor determines that the proposed publication contains confidential information, Sponsor may require the delay of publication for a period of time not to exceed 90 days and may require that any confidential information be removed from the publication. Sponsor may also require Physician to delay publication until any factual errors or inaccuracies in the publication are corrected.

DOCUMENTS (1):
  • Study Protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02040259/Prot_000.pdf